CLINICAL TRIAL: NCT04297059
Title: 2-year Intervention and 1-year Follow-up of a School-based Programme to Promote Healthy Behaviours and Prevent Childhood Obesity in Lebanese Children: the Healthier Kids - Ajyal Salima Study
Brief Title: The Ajyal Salima Longitudinal Study to Prevent Childhood Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NUT.NH.16
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Childhood Obesity
Keywords: BMI; Health policies; School health promotion; Intervention
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Implementation of Ajyal Salima intervention to promote healthy eating and encourage physical activity in Lebanese school-children.
  Interventions: Other: Ajyal Salima
- Control group (No Intervention): Group of students not receiving any intervention

INTERVENTIONS:
Other: Ajyal Salima — It comprises in class-activities, meetings with parents and improvement of school foodservice
  Arms: Intervention group

SUMMARY:
The study was carried out to determine the long-term effectiveness of a school-based intervention programme when implemented over 2 years and its sustained effect one year later.

ELIGIBILITY:
Inclusion Criteria:

Schoolchildren Aged 8-12 years

Exclusion Criteria:

* no exclusion criteria

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1239 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge score | 3 school years
  Change in the knowledge scores (the sum of correct answers) based on a scored questionnaire delivered during pre- and all post- assessment phases
Change in dietary habits | 3 school years
  Change in the percentage of children consuming sugary drinks, unhealthy and healthy snacks, fruits and vegetables/change in the percentage of children's physical activity frequency (self-reported in the questionnaires during pre- and all post- assessment phases)
Change in self-efficacy score | 3 school years
  Change in the self-efficacy scores (the sum of correct answers) based on a scored questionnaire delivered during pre- and all post- assessment phases
Change in Body Mass Index | 3 school years
  Change in mean BMIz scores (based on anthropometric measurements during pre- and post- assessment phases

IPD SHARING:
Plan to Share IPD: No